CLINICAL TRIAL: NCT01372436
Title: Caries Risk Assessment in Children and Adolescents in the Alpes Maritimes (France)
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: ARPSPBD2
Record Dates: First submitted 2008-04-22; First posted 2011-06-14 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-06

CONDITIONS: Children in School
Keywords: dental decay; DMFT; Individual Caries Risk; Risk factors
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: children in high-school
- 2: children in primary school

SUMMARY:
Identification of caries high risk subjects. Studying the relevance and the distribution of caries risk factors as defined by the HAS, and the part played by the zone of schooling (priority education area or not) Studying the interest of bacteriological tests using the technique of real-time PCR and the laser fluorescence device in the caries risk assessment Thanks to a prospective cohort study conducted over a period of 4 years on a representative sample of pupils and students chosen at random from the 360 primary schools and 89 high schools in the Alpes Maritimes (678 subjects).

DETAILED DESCRIPTION:
Main goal: Reducing social inequalities in dental health in the Alpes-Maritimes with the identification of high-risk subjects in order to implement effective preventive actions focused on people likely to benefit most from such actions.

Carrying out a prospective representative cohort, in schools, over a period of 4 years has the following objectives:

* To study the pattern of risk factors for tooth decay, as defined by the HAS, in the representative studied sample, and particularly to assess the part played by the zone of schooling (priority education area (low socio-economic) (PEA) or not).
* To evaluate, in a representative French sample, the relevance of the caries risk (CR) factors defined by the HAS based on an analysis of the foreign literature.
* To evaluate the interest of bacteriological tests using the technique of real-time PCR (Cario-analysis ®, Pierre Fabre Oral Care) in the assessment of CR, once the other risk factors are taken into account.
* To study the interest of using a laser fluorescence device (Diagnodent ® Pen, Kavo) compared to clinical examination alone, in the detection of caries which are difficult to diagnose(approximal caries or small enamel lesions) and its impact on the caries risk assessment.

Study Type: prospective cohort study. Population study: This study is conducted in 360 primary schools and 89 high-schools in the Alpes Maritimes (randomized study). They are divided into two strata (priority education area or not). Within each stratum and for each level of education (primary schools and high schools), schools are chosen at random on the corresponding list until the number of children needed in both the 1rst grade and the 5th grade is reached.

Pupils are followed by the investigators. Subjects Number: 678 (339 in 1rst grade and 339 in 5th grade proportionally divided into non-PEA and PEA).

Duration of follow-up: 4 years Frequency of visits: annual visits Oral health screening - clinical examination (probe and mirror) and with the new laser fluorescence device (DIAGNOdent ® pen, Kavo). Salivary Tests: bacteriological in real-time PCR (Cario-analysis ® Oral Care Pierre Fabre) and CRT Buffer ® Ivoclar Vivadent) Statistical analyses - Descriptive analyses and logistic regression models (dependent variable is the high caries risk (when CAODM36-CAODJ0 > or = 4)

ELIGIBILITY:
Inclusion Criteria:

- Enrolled in 1rst or 5th year (CP ou 6ème) at the beginning of the study

Exclusion criteria:

* Planning to change school or high school in the 4 years
* Refusing dental examination
* Refusing to chew the piece of paraffine

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children in primary or high-schools
Sampling Method: Probability Sample
Enrollment: 678 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
dental decay | every year

CONTACTS AND LOCATIONS:
Overall Officials: Michèle Muller Bolla, Pr, Principal Investigator — Odontologie - CHU de Nice
Locations (2):
- France (2):
  - Service d'Odontologie - Hôpital St Roch, Nice
  - Haute Autorité de Santé, Saint-Denis